CLINICAL TRIAL: NCT00765284
Title: Effect of Niaspan on Parameters of Reverse Cholesterol Transport and HDL-C Subclasses in Male Subjects With Low HDL-C Levels
Brief Title: Effect of Niaspan on Cholesterol in Men
Status: Completed | Type: Observational
Sponsor: KineMed (Industry)
Responsible Party: Drina Boban/ Clinical Studies Director, KineMed, Inc.
Other Study IDs: KM-12
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: HDL Cholesterol
Keywords: HDL; RCT; Cholesterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, urine, and blood samples will be taken and analyzed as part of the study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment: Ten subjects will be low HDL-C male volunteers who will receive aspirin and Niaspan
- Placebo: Five subjects will be low HDL-C male volunteers who will receive only aspirin.

SUMMARY:
To determine whether 8 weeks of Niaspan treatment increases cholesterol efflux in male subjects with low HDL-C cholesterol when compared to no treatment.

To determine whether 8 weeks of Niaspan treatment increases fecal cholesterol excretion when compared to no treatment.

To determine whether 8 weeks of Niaspan treatment increases the rate of global reverse cholesterol transport when compared to no treatment.

DETAILED DESCRIPTION:
This will be a single center, open-label, randomized, mechanism of action study consisting of 8 weeks of active treatment preceded by a screening phase from one to 8 weeks and a baseline measurement of parameters of reverse cholesterol transport for 10 days. The population for this trial is 15 non-diabetic men aged 18-70 years. Ten subjects will be low HDL-C male volunteers who will receive aspirin and Niaspan and five subjects will be low HDL-C male volunteers who will receive only aspirin.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following criteria at the Screening Visit will be eligible to participate:

* Provide written informed consent
* Male
* Age 18 to 70 years
* BMI 18.5-40 kg/m2
* HDL-C values <40 mg/dL
* Triglyceride value 150-500 mg/dL.
* Good health based on medical history, physical examination and laboratory safety tests performed at the screening visit or prior to initial dose of study medication.
* No clinically significant abnormality on ECG performed at the screening visit or prior to initial dose of study medication.
* Non-smoker and no other use of nicotine containing products for at least 6 months and does not plan to begin smoking during the course of the study.
* Dietary or nutritional remedies including plant sterol containing products (i.e. Benecol, SmartBalance, etc) of any sort for at least 2 weeks prior to and throughout the study.
* Willing to avoid the use of lipid modifying medications (excluding statins) such as the fibrates, cholestyramine, fish oil, and ezetimibe within 8 weeks prior to and during the study.
* Avoidance of extreme change of physical activity from screening through the follow-up period.

Exclusion Criteria:

Subjects are excluded from participation in the study if any of the following criteria apply:

* History of intolerance to Niacin or Niaspan.
* Treatment with Niacin or Niaspan in the past 3 months (Multivitamin use with non-pharmacologic doses of Niacin - less than 500mg per day - is allowed).
* History of stroke, chronic seizures, or major neurological disorder.
* Significant emotional problems or a history of clinically significant psychiatric disorder.
* Bleeding diathesis or intolerance to aspirin.
* Anemia as defined as a hematocrit < 25%.
* History of gastritis, bleeding gastric or duodenal ulcers.
* History Type 1 or Type 2 diabetes, or fasting plasma glucose >125 mg/dL at screening or 75 gm OGTT with 2 hour glucose >140mg/dL.
* History of illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk through participation.
* History of ileal bypass, gastric bypass, or other condition associated with malabsorption.
* Abnormal thyroid function tests.
* AST or ALT > 1.5x the upper limit of normal.
* Active or recent gastrointestinal condition such as gastroenteritis, irritable bowel syndrome, chronic constipation, or diarrhea which may affect bowel movements.
* History of plant sterol storage disease or a history of intolerance to plant sterols or plant sterol containing products.
* History of neoplastic disease (i.e. leukemia, lymphoma, malignant melanoma), or myeloproliferative disease, regardless of the time since treatment. Exceptions include adequately treated non-melanomatous skin carcinoma, and other malignancies that may have been treated successfully >10 years prior to the screening visit with no evidence of recurrence.
* Excessive alcohol consumption defined as > three glasses of alcoholic beverages or distilled spirits per day. *** Must avoid excessive alcohol consumption throughout study.
* Currently using psyllium or other fiber based laxatives, phytosterol margarines, and/or over the counter (OTC) treatments that are known to affect serum lipids and has NOT been treated with a stable regimen for > 6 weeks prior to screening (Visit 1) or the subject DOES NOT agree to continue this regimen for the duration of the clinical trial.
* Regular user of illicit drugs or history of drug abuse (including alcohol) within the previous 2 years.
* Use of anabolic agents.
* Any condition or therapy which, in the opinion of the investigator, poses a risk to the subject
* Use of any investigational drug within 30 days before screening

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study will include a total of 15 subjects, non-diabetic men with low HDL-C, defined as <40 mg/dL. Subjects will be aged 18 to 70 years and have a BMI between 18.5-40 kg/m2.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2007-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To determine whether 8 weeks of Niaspan treatment increases the following: cholesterol efflux, fecal cholesterol excretion, and the rate of global reverse cholesterol transport, in male subjects with low HDL-C cholesterol when compared to no treatment. | 8 weeks

SECONDARY OUTCOMES:
To measure the longitudinal effects of 8 weeks of Niaspan treatment on percent change in concentration of specific HDL-C sub-fractions when compared to no treatment. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Scott Turner, PhD, Study Director — KineMed, Inc.
Locations (1):
- Diabetes and Glandular Research Associates, San Antonio, Texas, United States